CLINICAL TRIAL: NCT00278499
Title: Epidemiology of HIV-1 and Other Sexually Transmitted Infections in Honghe Prefecture, Yunnan Province, China
Brief Title: Prevalence of HIV and Other Sexually Transmitted Infections Among Female Sex Workers and Miners in Honghe Prefecture, Yunnan Province, China
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Other Study IDs: CIPRA CH 005; CIPRA Project 1
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2011-01

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Cross-Sectional Studies; Surveys and Questionnaires; Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Female sex workers
  Interventions: Behavioral: Cross-sectional surveys
- 2: Female sex workers' clients (miners)
  Interventions: Behavioral: Questionnaire/counseling

INTERVENTIONS:
Behavioral: Cross-sectional surveys — Cross-sectional surveys will occur at study entry, Month 6, and Month 12. Every fourth participant enrolled in the FSW cross-sectional survey, all FSWs found to be HIV infected, and all FSWs who are intravenous drug users will participate in a substudy lasting 12 months.
  Groups: 1
Behavioral: Questionnaire/counseling — An initial questionnaire and counseling will occur once in addition to post-test counseling.
  Groups: 2

SUMMARY:
The purpose of this study is to collect data on the HIV strains currently circulating among female sex workers (FSWs) and their clients. In addition, this study will identify potential participants for future studies.

DETAILED DESCRIPTION:
The overwhelming majority of HIV/AIDS patients live in the developing world. The rate of HIV infection in China has been consistently and steadily increasing over the past few years. Commercial sex workers and their clients are at highest risk for HIV infection and transmission. Yunnan Province is reported to be home to about half of China's HIV infected population. Honghe Prefecture accounts for 14% of the total reported HIV infections in Yunnan Province. Even though the incidence of HIV is important in tracking the HIV epidemic, there are little data on HIV incidence among FSWs in China. Estimates of HIV incidence are essential for optimally monitoring the HIV epidemic, knowing where to focus prevention efforts, and evaluating the success of vaccines and other prevention strategies. The purpose of this study is to estimate the incidence of and risk factors for HIV infection among FSWs and miners in Honghe Prefecture, Yunnan Province, China. In addition, this study will identify and describe the different HIV clades currently circulating among FSWs and miners. Four cross-sectional surveys will be conducted: three among FSWs and one among miners. In addition, a 12-month cohort study will be conducted among a subgroup of FSWs enrolled in the baseline cross-sectional survey in Kaiyuan City, Honghe Prefecture, Yunnan Province, China.

FSWs will complete cross-sectional surveys at study entry, Month 6, and Month 12. FSWs will complete two study visits: one to complete the survey and another to receive test results and participate in post-test counseling. Physical and gynecologic exams and blood collection will occur at both study visits. Each survey will include general participant information and sexual activity and drug use habits.

Pre-test counseling will be provided to all FSWs; those who elect to donate specimens for laboratory testing will have an additional appointment within 6 weeks of donation to receive test results and post-test counseling. Multiple counseling sessions may be provided to some participants based on their individual needs. FSWs found to be either infected with HIV or another sexually transmitted disease (STD) will be referred for further medical evaluation and treatment.

Every fourth participant enrolled in the FSW cross-sectional survey, all FSWs found to be HIV infected, and all FSWs who are intravenous drug users will participate in a substudy lasting 12 months. Study staff will contact each participant once a month for 12 months and ask them for location information and about their current behaviors.

Participants enrolled as FSW clients (miners) will participate in two study visits. The first visit will include completing a questionnaire and counseling. The second study visit will include post-test counseling to inform participants of their test results and will occur about one month after the first visit. A physical exam and blood and urine collection will occur at both visits.

ELIGIBILITY:
Inclusion Criteria for FSWs Completing Cross-sectional Survey:

* Self-reported to have sold sex for money within the 3 months prior to study entry
* Works at one of the study sites

Inclusion Criteria for FSW Cohort Study:

* Participated in the baseline cross-sectional survey in Kaiyuan City, Honghe Prefecture, Yunnan Province, China
* Willing to provide updated contact information (and a cell phone number, if available)
* Willing to be contacted by study staff once a month for 12 consecutive months

Inclusion Criteria for FSW Client (Miner) Study:

* Male
* Works at one of the selected mine sites

Inclusion Criteria for All Participants:

* Parent or guardian willing to provide informed consent, if applicable

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Female sex workers and their clients in Hinghe Prefecture, Yunnan Province, China
Sampling Method: Non-Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2006-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Incidence of HIV-1 infection in FSWs and mine workers | Throughout study
Risk factors for HIV-1 infection including, but not limited to injection drug use, STIs, and unprotected sex among FSWs and mine workers separately | Throughout study

SECONDARY OUTCOMES:
Prevalence of HIV-1 infection and selected STIs | Throughout study
HIV/STI related knowledge, attitudes, and risk behaviors in FSWs and mine workers separately | Throughout study
HIV-1 viral subtypes in FSWs and mine workers separately | Throughout study
FSW migration patterns in a sub-cohort of FSWs | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ning Wang, MD, PhD, Principal Investigator — Chinese Center for Disease Control and Prevention, National Center for AIDS/STD Prevention and Control; Zhongmin Yang, MD, Principal Investigator — Chinese Center for Disease Control and Prevention, National Center for AIDS/STD Prevention and Control
Locations (2):
- China (2):
  - Gejiu CDC, Honghe Prefecture, Yunnan Province, Kunming, Yunnan
  - Kaiyuan CDC, Honghe, Kunming, Yunnan

REFERENCES:
- [Background] Anderson AF, Qingsi Z, Hua X, Jianfeng B. China's floating population and the potential for HIV transmission: a social-behavioural perspective. AIDS Care. 2003 Apr;15(2):177-85. doi: 10.1080/0954012031000068326. PMID 12856339
- [Background] Chen XS, Yin YP, Liang GJ, Gong XD, Li HS, Poumerol G, Thuy N, Shi MQ, Yu YH. Sexually transmitted infections among female sex workers in Yunnan, China. AIDS Patient Care STDS. 2005 Dec;19(12):853-60. doi: 10.1089/apc.2005.19.853. PMID 16375618
- [Background] Ding Y, Detels R, Zhao Z, Zhu Y, Zhu G, Zhang B, Shen T, Xue X. HIV infection and sexually transmitted diseases in female commercial sex workers in China. J Acquir Immune Defic Syndr. 2005 Mar 1;38(3):314-9. PMID 15735451
- [Background] Tucker JD, Henderson GE, Wang TF, Huang YY, Parish W, Pan SM, Chen XS, Cohen MS. Surplus men, sex work, and the spread of HIV in China. AIDS. 2005 Mar 24;19(6):539-47. doi: 10.1097/01.aids.0000163929.84154.87. PMID 15802971
- [Background] Zhao R, Gao H, Shi X, Tucker JD, Yang Z, Min X, Qian H, Duan Q, Wang N. Sexually transmitted disease/HIV and heterosexual risk among miners in townships of Yunnan Province, China. AIDS Patient Care STDS. 2005 Dec;19(12):848-52. doi: 10.1089/apc.2005.19.848. PMID 16375617